CLINICAL TRIAL: NCT04991428
Title: Mechanism of Action of Transcranial Direct Current Stimulation in Neurofibromatosis Type 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Dr Shruti Garg, Clinical Senior Lecturer, University of Manchester
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 18/NW/0762
Record Dates: First submitted 2021-07-27; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Neurofibromatosis 1
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Single-blind cross over experimental trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active trancranial direct current stimulation (Experimental): Active stimulation for 15 minutes
  Interventions: Other: Transcranial direct current stimulation
- Sham stimulation (Sham Comparator): Similar set-up but no actual stimulation
  Interventions: Other: Transcranial direct current stimulation

INTERVENTIONS:
Other: Transcranial direct current stimulation — tDCS is a form of non-invasive brain stimulation. tDCS is an established research tool for non-invasive modulation of neuroplasticity. It uses low-intensity DC currents to modulate spontaneous neuronal network activity by altering the resting membrane potential. Anodal tDCS has been shown to increase cortical excitability, reduce regional levels of GABA enhance LTP and synaptic plasticity.

SUMMARY:
Intellectual impairment, particularly working memory deficits are a significant cause of morbidity in children with Neurofibromatosis type (NF1) with long-term implications on academic and occupational functioning. Whilst significant discoveries have been made in Nf1 animal models in trying to find treatments for these conditions, human translational studies have not been successful. This mechanistic experimental study will investigate the neural mechanisms underlying working memory deficits in NF1. In particular, we will investigate how individual differences in inhibitory neurotransmitter GABA relate to performance on working memory tests. Further, we will investigate the use of a novel, experimental intervention called transcranial Direct Current Stimulation (tDCS);known to modulate GABA. Using a randomized, crossover design in a cohort of 30 adolescents aged 11-17 years, we will apply real or sham tDCS to the dorsolateral prefrontal cortex (DLPFC). State-of-art real time imaging techniques such as Magnetic Resonance Spectroscopy (MRS) and task based functional MRI (fMRI) will be used to investigate the effect of tDCS on GABA concentration, changes in functional plasticity and working memory. We expect that results from this study will help elucidate the neural mechanisms underlying working memory deficits in people with NF1 and show biologic activity for a novel, low-cost intervention that can be used for cognitive remediation in NF1. This kind of focused mechanism trial method is a highly promising approach to understanding the complex neural system pathology in a multifactorial neurodevelopmental condition like NF1.

ELIGIBILITY:
Inclusion Criteria:

1. Meets National Institute of Health NF1 diagnostic criteria
2. Children aged 11-17 years
3. Written informed consent/assent

Exclusion Criteria:

1. No history of intracranial pathology other than asymptomatic optic pathway glioma or other asymptomatic and untreated NF1-associated white matter lesion
2. No history of epilepsy or any major mental illness
3. No MRI contraindications.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Corsi Block task | immediately after the intervention
  memory span task

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manchester, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Collected data will be available to share after publication of study findings
Supporting Information: Study Protocol
Time Frame: The data will be made available upon request.